CLINICAL TRIAL: NCT05144113
Title: FES-Rowing: Preventing the Secondary Conditions of Paralysis Through Vigorous Exercise
Status: Completed | Type: Observational
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, J. Andrew Taylor, Associate Professor, Spaulding Rehabilitation Hospital
Other Study IDs: 2020P003132; 1R41HD102267-01A1 (NIH)
Record Dates: First submitted 2021-08-04; First posted 2021-12-03 (Actual); Results first posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Paralysis, Legs
MeSH Terms: conditions — Paraplegia | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Current FES-Row Subjects: To determine user needs we will survey 10 subjects that are currently participating in FES-row training to discover their motivations, preferences and challenges pertaining to participation in physical activity in general and FES-rowing.
  Interventions: Behavioral: Survey subjects to discover their motivations, preferences and challenges pertaining to participation in physical activity in general and FES-rowing.
- Non-FES-Row Subjects: To determine user needs we will survey 10 subjects that have never participated in FES-row training to discover their motivations, preferences and challenges pertaining to participation in physical activity in general and FES-rowing.
  Interventions: Behavioral: Survey subjects to discover their motivations, preferences and challenges pertaining to participation in physical activity in general and FES-rowing.

INTERVENTIONS:
Behavioral: Survey subjects to discover their motivations, preferences and challenges pertaining to participation in physical activity in general and FES-rowing. — The following questionnaires will be answered by subjects:
  Questionnaires:
  Barriers to Physical Activity Questionnaire for People with Mobility Impairments (BPAQ-MI): measures barriers to physical activity across the intrapersonal and interpersonal domains.
  Physical Activity and Disability Survey (PADS): measures physical activity for people with chronic neurological conditions.
  Demographic and Mobility Questionnaire: Important information to inform on user and design needs and potential market for at home FES-row system.
  Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0)-(FES-row participants only): measures satisfaction with current FES-row system used in the ExPD Program.

SUMMARY:
Over the past ten years, the Cardiovascular Research Laboratory at Spaulding has refined a unique form of exercise for those with spinal cord injuries (SCI). Functional Electrical Stimulation Row Training (FESRT) couples volitional arm and electrically controlled leg exercise, resulting in the benefits of large muscle mass exercise. Despite the success of the FES-rowing Program at Spaulding, FES-rowing systems have not yet evolved beyond research prototypes, and ours is the only program in the US where FES-rowing is available. A new design is critically needed to enable people with paralysis to participate in FES rowing in their own homes, which we believe will maximize both the health and commercial impacts of FES-rowing.

DETAILED DESCRIPTION:
The purpose of this observational study is to gain insights into user needs, and market perception of physical activity and FES-rowing to further develop a new, home-based FES-rowing system that meets the needs of people with paralysis. We will enroll a total of 20 subjects, male and female, 18 years and older with lower-limb paralysis who use a wheelchair as their primary means of mobility. Ten subjects will be current FES-rowing participants (especially those doing FES-rowing at home) and 10 subjects will be non-participants. To determine user needs we will survey prospective customers to discover their motivations, preferences and challenges pertaining to participation in physical activity in general and FES-rowing.

Questionnaires:

Barriers to Physical Activity Questionnaire for People with Mobility Impairments (BPAQ-MI): measures barriers to physical activity across the intrapersonal and interpersonal domains.

Physical Activity and Disability Survey (PADS): measures physical activity for people with chronic neurological conditions.

Demographic and Mobility Questionnaire: Important information to inform on user and design needs and potential market for at home FES-row system.

Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0)-(FES-row participants only): measures satisfaction with current FES-row system used in the ExPD Program.

ELIGIBILITY:
* male and female,
* 18 years of age and older
* lower-limb paralysis who use a wheelchair as their primary means of mobility.

Exclusion Criteria:

* Under 18 years of age
* no lower-limb paralysis
* People who do not use a wheelchair as their primary means of mobility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 subjects, male and female, 18 years and older with lower-limb paralysis who use a wheelchair as their primary means of mobility. Ten subjects will be current FES-rowing participants (especially those doing FES-rowing at home) and 10 subjects will be non-participants.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Hospital Cambridge, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient department of Rehabilitation Hospital
Groups:
- Current FES-Row Subjects: To determine user needs we will survey 10 subjects that are currently participating in FES-row training to discover their motivations, preferences and challenges pertaining to participation in physical activity in general and FES-rowing.
  Survey subjects to discover their motivations, preferences and challenges pertaining to participation in physical activity in general and FES-rowing.: The following questionnaires will be answered by subjects:
  Questionnaires:
  Barriers to Physical Activity Questionnaire for People with Mobility Impairments (BPAQ-MI): measures barriers to physical activity across the intrapersonal, interpersonal, organizational, and community domains.
  Physical Activity and Disability Survey (PADS): measures physical activity for people with chronic neurological conditions.
  Demographic and Mobility Questionnaire: Important information to inform on user and design needs and potential market for at home FES-row system.
  Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0)-(FES-row participants only): measures satisfaction with current FES-row system used in the ExPD Program.
- Non-FES-Row Subjects: To determine user needs we will survey 10 subjects that have never participated in FES-row training to discover their motivations, preferences and challenges pertaining to participation in physical activity in general and FES-rowing.
  Survey subjects to discover their motivations, preferences and challenges pertaining to participation in physical activity in general and FES-rowing.: The following questionnaires will be answered by subjects:
  Questionnaires:
  Barriers to Physical Activity Questionnaire for People with Mobility Impairments (BPAQ-MI): measures barriers to physical activity across the intrapersonal, interpersonal, organizational, and community domains.
  Physical Activity and Disability Survey (PADS): measures physical activity for people with chronic neurological conditions.
  Demographic and Mobility Questionnaire: Important information to inform on user and design needs and potential market for at home FES-row system.
  Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0)-(FES-row participants only): measures satisfaction with current FES-row system used in the ExPD Program.
Period: Overall Study
Arm/Group | Current FES-Row Subjects | Non-FES-Row Subjects
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- FES-row Training: 10 subjects, male and female, 18 years and older with lower limb paralysis who use a wheelchair as their primary means of mobility and are currently participating in FES-row training
- Non-FES-row Training: 10 subjects, male and female, 18 years and older with lower limb paralysis who use a wheelchair as their primary means of mobility and are not currently participating in FES-row training
- Total: Total of all reporting groups
Arm/Group | FES-row Training | Non-FES-row Training | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (17.0) | 43.1 (13.7) | 44.5 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 9 | 7 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Barriers to Physical Activity Questionnaire for People With Mobility Impairments (BPAQ-MI)
Description: measures barriers to physical activity across the intrapersonal (health and beliefs/attitudes) and interpersonal (friends and family) domains. Minimum score is 0 (not a barrier at all), and larger scores up to a maximum domain score of 5 indicate bigger barriers to physical activity.
Time Frame: baseline
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Current FES-Row Subjects: Subjects who were currently training with functional electrical stimulation (FES) rowing.
- Non FES-Row Subjects: Subjects who were not a part of the functional electrical stimulation (FES) row training program.
Arm/Group | Current FES-Row Subjects | Non FES-Row Subjects
Number analyzed (Participants) | 10 | 10
units on a scale
  Intrapersonal Domain: Health | 0.66 (0.18) | 1.24 (0.20)
  Intrapersonal Domain: Beliefs/Attitudes | 0.22 (0.13) | 0.06 (0.05)
  Interpersonal Domain: Friends | 0.83 (0.18) | 1.56 (0.44)
  Interpersonal Domain: Family | 0.96 (0.27) | 1.35 (0.49)

2. Primary Outcome: Barriers to Physical Activity and Disability Survey (BPAD-S)
Description: measures barriers to physical activity for people with chronic neurological conditions by asking each subject to endorse/deny (i.e., yes/no) experiencing 19 unique barriers. Number of subject endorsements ("yes") of each barrier per group (Current FES-Row vs. Non FES-Row) are reported. Thus, the sum of the rows will not equal the number of participants analyzed, since subject could endorse experiencing up to 19 barriers.
Time Frame: baseline
Population: Two subjects in the Current FES-Row group did not complete the BPAD-S and were therefore excluded from analysis (n=8 FES-Row, n=10 non FES-Row).
Measure: Count of Participants; unit: Participants
Arm/Group | Current FES-Row Subjects | Non FES-Row Subjects
Number analyzed (Participants) | 8 | 10
Participants
  Barrier: cost of exercise program | 5 | 3
  Barrier: lack of transportation | 2 | 3
  Barrier: lack of time | 4 | 2
  Barrier: lack of interest | 1 | 0
  Barrier: lack of energy | 2 | 3
  Barrier: lack of motivation | 2 | 2
  Barrier: lack of support from friends or family to exercise | 1 | 0
  Barrier: lack of personal care attendant who will help me exercise | 3 | 1
  Barrier: lack of accessible facility | 3 | 4
  Barrier: exercise is boring or monotonous | 0 | 1
  Barrier: exercise will not improve my condition | 0 | 1
  Barrier: exercise will make my condition worse | 0 | 1
  Barrier: exercising is too difficult | 0 | 1
  Barrier: don't know how to exercise | 1 | 2
  Barrier: don't know where to exercise | 1 | 3
  Barrier: health concerns prevent me from exercising | 2 | 3
  Barrier: pain prevents me from exercising | 3 | 4
  Barrier: I am too old to exercise | 0 | 0
  Barrier: feel uncomfortable or self-conscious in a fitness center | 2 | 0

3. Primary Outcome: Demographic and Mobility Questionnaire: Clinical Diagnosis Causing Paralysis
Description: important information to inform on user and design needs and potential market for at home FES-row system.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | FES-row Training | Non-FES-row Training
Number analyzed (Participants) | 10 | 10
Participants
  Cerebral palsy | 0 | 1
  Multiple schlerosis | 1 | 3
  Spinal cord injury | 9 | 5
  Spina bifida | 0 | 1

4. Primary Outcome: Demographic and Mobility Questionnaire: Type of Wheelchair Primarily Used
Description: important information to inform on user and design needs and potential market for at home FES-row system.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Current FES-Row Subjects | Non FES-Row Subjects
Number analyzed (Participants) | 10 | 10
Participants
  Manual wheelchair | 7 | 8
  Power wheelchair | 3 | 2

5. Primary Outcome: Quebec User Evaluation of Satisfaction With Assistive Technology (QUEST 2.0)
Description: (FES-row participants only): measures satisfaction with current FES-row system used in the ExPD Program. Minimum score is 0 (least satisfied), maximum score is 5 (most satisfied).
Time Frame: baseline
Population: Only subjects who were currently training with functional electrical stimulation (FES) rowing.
Measure: Mean (Standard Error); unit: score on scale
Groups:
- Current FES-Row Subjects: FES-row training
Arm/Group | Current FES-Row Subjects
Number analyzed (Participants) | 10
score on scale | 4.45 (0.16)

ADVERSE EVENTS:
Time Frame: 1 Day, single visit
Arm/Group | Current FES-Row Subjects | Non-FES-Row Subjects
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT05144113/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT05144113/SAP_001.pdf